CLINICAL TRIAL: NCT02917512
Title: A Multicenter, Placebo Controlled, Restasis® Referenced, Randomized, Double Blind, Phase II Study to Evaluate the Efficacy and Safety of HU00701/HU007 Eye Drops in Patients With Dry Eye Syndrome
Brief Title: Efficacy and Safety Study of HU00701/HU007 Eye Drops in Patients With Dry Eye Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HU-007_P2
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- HU00701 (Experimental): HU00701(Cyclosporine 0.01% + 3% trehalose)
  1 drop b.i.d at 12 hour interval for 12 weeks
  Interventions: Drug: HU00701
- HU007 (Experimental): HU007(Cyclosporine 0.02% + 3% trehalose)
  1 drop b.i.d at 12 hour interval for 12 weeks
  Interventions: Drug: HU007
- Restasis (Active Comparator): Restasis(Cyclosporine 0.05%)
  1 drop b.i.d at 12 hour interval for 12 weeks
  Interventions: Drug: Restasis
- Placebo(without main component) (Placebo Comparator): Placebo
  1 drop b.i.d at 12 hour interval for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HU00701 — Cyclosporine 0.01% + 3% trehalose
  Arms: HU00701
Drug: HU007 — Cyclosporine 0.02% + 3% trehalose
  Arms: HU007
Drug: Restasis — Cyclosporine 0.05%
  Arms: Restasis
Drug: Placebo — Vehicle
  Arms: Placebo(without main component)

SUMMARY:
A multicenter, Placebo controlled, Restasis® referenced, Randomized, Double blind, Phase II Study to Evaluate the Efficacy and Safety of HU00701/HU007 Eye Drops in Adult Patients with Dry Eye Syndrome

ELIGIBILITY:
Inclusion Criteria:

* age over 19
* Corneal staining score(Oxford grading) > 2 or Schirmer test < 10mm/5min (If Schirmer test = 0mm/5min, Nasal stimulation schirmer test > 3mm/5min)
* Volunteer who went through menopause more than 1 years ago before screening or has surgical menopause
* Volunteer who has negative result of pregnancy test or use effective contraception

Exclusion Criteria:

* Current or recent patients used dry eye syndrome medications (topical or systemic) that may affect the status
* The patients with systemic or ocular disorders affected the test result
* Being treated with systemic steroid
* Wearing contact lenses within 3 days of screening visit
* Pregnancy or Breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
change from Baseline of Corneal staining score - Oxford grading | Week 12

SECONDARY OUTCOMES:
change from Baseline of Corneal staining score - Oxford grading | Week 4, 8
change from Baseline of Strip meniscometry assessment | Week 4, 8, 12
change from Baseline of Tear film break-up time | Week 4, 8, 12
change from Baseline of Standard patient evaluation of eye dryness questionnaire | Week 4, 8, 12

CONTACTS AND LOCATIONS:
Overall Officials: Seung-il Baek, Study Director — Huons Co., Ltd.
Locations (1):
- Huons, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shin J, Rho CR, Hyon JY, Chung TY, Yoon KC, Joo CK. A Randomized, Placebo-Controlled Phase II Clinical Trial of 0.01% or 0.02% Cyclosporin A with 3% Trehalose in Patients with Dry Eye Disease. J Ocul Pharmacol Ther. 2021 Jan-Feb;37(1):4-11. doi: 10.1089/jop.2020.0104. PMID 33449860